CLINICAL TRIAL: NCT02134340
Title: A Phase 1a, Multi-centre, Open-label, Non-randomized Study to Assess the Safety, Biodistribution and Tumour Uptake of [I-124]-CPD-1028 Injection
Brief Title: A Safety and Biodistribution Study of [I-124]-CPD-1028 Injection in Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Probe Development and Commercialization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPD1028-01
Record Dates: First submitted 2014-04-14; First posted 2014-05-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: IGF1R
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [I-124]-CPD-1028 PET/CT (Experimental): Administration of [I-124]-CPD-1028 Injection followed by a maximum of 3 PET/CT imaging sessions.
  A pre-targeting dose of CPD-1061 may be given prior to injection of [I-124]-CPD-1028.
  Interventions: Drug: [I-124]-CPD-1028 Injection; Biological: CPD-1061

INTERVENTIONS:
Drug: [I-124]-CPD-1028 Injection — A single intravenous dose of [I-124]-CPD-1028 Injection will be given at Visit 2 (within 21 days of screening Visit 1), and may be followed by whole body PET/CT imaging approximately 3 hours post-injection. PET/CT imaging will occur at Visit 3 (2-3 days after Visit 2) and Visit 4 (5-7 days after Visit 2). PET/CT imaging may also occur at Visit 5 (16-18 days after Visit 2). Visit 6 (28 +/- 2 days after Visit 2) is a follow-up telephone call for a post-treatment safety assessment. At Visits 2-5, whole body biodistribution and tumour uptake will be assessed. At all visits, safety will be assessed.
Biological: CPD-1061 — [Optional] An intravenous dose of 0.4, 1.4 or 6 mg/kg of body weight of CPD-1061 may be given 1-2 hours prior to injection of [I-124]-CPD-1028 at Visit 2. The decision to use CPD-1061 and the dose amount is based on an adaptive design and is dependent on interim reviews of imaging data.

SUMMARY:
The purpose of the study is to evaluate the safety and biodistribution of [I-124]-CPD-1028 Injection in cancer patients with solid tumours.

DETAILED DESCRIPTION:
Up to 18 adult participants will be enrolled in this Phase 1a study to evaluate the safety and biodistribution of [I-124]-CPD-1028 Injection in patients with Insulin-like Growth Factor-1R (IGF-1R) upregulated solid tumours. All eligible subjects who have given written informed consent and qualify based on the study's inclusion/exclusion criteria will be enrolled in the study. Each enrolled subject will take part in six visits consisting of a screening visit, an Investigational Product administration visit, 3 assessment visits involving 2-3 Positron Emission Tomography/Computed Tomography (PET/CT) scans, and a follow-up safety telephone call. At Visit 2, subjects will start a course of treatment to protect the thyroid from radioactivity and may receive a pre-targeting dose of an additional investigational agent, CPD-1061.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old with life expectancy > 12 weeks with confirmed metastatic or unresectable malignancy
2. Patients must have progressed after at least first-line chemotherapy and have an Eastern Cooperative Oncology Group (ECOG) status of 0, 1 or 2.
3. All patients must have archival tumour samples available and must have verification of IGF-1R expression.
4. Patients must have adequate organ and marrow function, vital signs and ECG.
5. Females of childbearing potential must not be pregnant and both males and females must use adequate forms of contraception.
6. Signed informed consent form
7. Subject must be compliant and have a high probability of completing the study.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from previous treatment.
2. Patients who have received a therapeutic radiopharmaceutical in the past year or who are currently receiving any other investigational agents.
3. Previous treatment with IGF-1R inhibitors.
4. Patients who are currently taking antithyroid medications and lithium or potassium sparing diuretics.
5. Subjects with known or suspected allergies or contraindications to the investigational agents and iodine
6. Subjects with uncontrolled intercurrent illness
7. Female subjects who are pregnant, planning to become pregnant or are lactating and/or breast-feeding.
8. Patients with diabetes requiring therapy unless controlled through diet or metformin.
9. Subjects who are undergoing monitoring of occupational ionising radiation exposure.
10. Subjects with hypothyroidism requiring thyroid supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evaluate safety of [I-124]-CPD-1028 Injection | Up to 30 days
  The safety of [I-124]-CPD-1028 Injection will be assessed for up to 30 days post injection by measuring the occurrence of adverse events and changes from baseline in physical examination, clinical laboratory parameters, electrocardiogram recordings, and vital signs (blood pressure, heart rate, body temperature, respiratory rate and oxygen saturation).
Obtain preliminary biodistribution data for [I-124]-CPD-1028 | Up to 18 days
  Biodistribution data will be assessed by quantitative analysis of imaging scans taken 2-3 days and 5-7 days post injection by (1) measuring tumour uptake and background tissue levels in selected regions of interest on whole body images and (2) determining if suitable quantitative imaging metrics can be identified.

SECONDARY OUTCOMES:
Measure blood and plasma clearance of [I-124]-CPD-1028 and levels of free [I-124]-Iodide | Up to 18 days
  Blood and plasma clearance of [I-124]-CPD-1028 and levels of free [I-124]-iodide will be assessed by analysis of blood and plasma samples taken up to 18 days post-injection.
Compare [I-124]-CPD-1028 uptake in tumours to IGF-1R expression | Up to 18 days
  [I-124]-CPD-1028 PET/CT images taken up to 18 days post-injection will be compared to immunohistochemistry staining scores of IGF-1R on previously obtained tumour samples.
Compare [I-124]-CPD-1028 PET/CT images to other imaging modalities | Up to 18 days
  [I-124]-CPD-1028 PET/CT images taken up to 18 days post-injection will be visually (qualitatively) compared to previously obtained CT and/or MRI images.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Burak, PhD, Study Director — Centre for Probe Development and Commercialization
Locations (4):
- Canada (4):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Science Centre - Odette Cancer Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario